CLINICAL TRIAL: NCT00715923
Title: CTSA Utility of Modified Consent Forms in Clinical Research: Fraga Tea Study
Brief Title: Modified Consent Form Utility
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: funding
Sponsor: University of California, Davis (Other)
Collaborators: National Center for Research Resources (NCRR) (NIH)
Responsible Party: Principal Investigator, Alexander A. Kon, MD, Professor, University of California, Davis
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 200715802
Record Dates: First submitted 2008-07-11; First posted 2008-07-15 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Healthy
Keywords: informed consent document; ethics

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Modified consent form
  Interventions: Other: Modified consent form
- 2 (Active Comparator): Standard consent form
  Interventions: Other: Standard consent form

INTERVENTIONS:
Other: Modified consent form — modified consent form used
  Arms: 1
Other: Standard consent form — standard consent form used
  Arms: 2

SUMMARY:
Subjects enrolling into a nutrition study of the effects of tea on fat absorption will be randomized to receive either a standard informed consent document or a modified document that is shorter and more easily understood than the standard document. The hypothesis is that using a shorter form that is more easily understood and more visually simple will lead to greater subject satisfaction in the consent process and will not compromise subject comprehension of key study aspects. Consent for study inclusion has been waived by the IRB because informing subjects of the nature and process of the study would likely affect the findings, and both the standard and modified consent forms were approved for use in the nutrition study.

ELIGIBILITY:
Inclusion Criteria:

* participation in parent study, English speaking

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2007-11; Primary Completion 2008-09 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Subject satisfaction | close of parent study

CONTACTS AND LOCATIONS:
Overall Officials: Alexander A Kon, MD, Principal Investigator — University of California, Davis
Locations (1):
- University of California Davis, Sacramento, California, United States